CLINICAL TRIAL: NCT06043973
Title: A Prospective Single-center, Single-arm Clinical Study of Almonertinib Combined With Anlotinib as First-line Treatment for Advanced Non-small Cell Lung Cancer With EGFR Sensitive Mutation and TP53 Mutation
Brief Title: Almonertinib Combined With Anlotinib as First-line Treatment for Advanced Non-small Cell Lung Cance
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2023(090)
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: almonertinib; anlotinib; EGFR mutation; TP53 mutation; advanced non-small cell lung cancer
MeSH Terms: interventions — aumolertinib; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- almonertinib plus anlotinib (Experimental): The specific treatment regimen is as follows: Non-squamous NSCLC: almonertinib (110 mg/d) plus anlotinib (12mg/d) is started on the first day of each treatment cycle and administered every three weeks until disease progression or intolerable toxicity. Anlotinib was given for two weeks, followed by one week off.
  Interventions: Drug: almonertinib

INTERVENTIONS:
Drug: almonertinib — The specific treatment regimen is as follows: Non-squamous NSCLC: almonertinib (110 mg/d) plus anlotinib (12mg/d) is started on the first day of each treatment cycle and administered every three weeks until disease progression or intolerable toxicity. Anlotinib was given for two weeks, followed by one week off.
  Other Names: Anlotinib

SUMMARY:
To evaluate the efficacy and safety of almonertinib plus anlotinib as first-line treatment for advanced non-small cell lung cancer with EGFR sensitive mutation and TP53 mutation.

This study is an exploratory single-arm study. The specific treatment regimen is as follows: Non-squamous NSCLC: almonertinib (110 mg/d) plus anlotinib (12mg/d) is started on the first day of each treatment cycle and administered every three weeks until disease progression or intolerable toxicity. Anlotinib was given for two weeks, followed by one week off.

Patients are assessed for measurable disease at baseline, 6 weeks, 12 weeks after starting treatment, and every 9 weeks thereafter according to RECIST 1.1 criteria during the treatment period until disease progression or intolerable toxicity withdrawal. Following discontinuation of treatment, subjects are followed for survival status every 3 months until death. Subject safety was assessed during treatment according to NCI CTCAE Version 4.0 criteria. Subjects who experience an AE should be followed until the AE returns to baseline. The primary endpoints is Progression-free survival (PFS) . Secondary endpoints include objective response rate (ORR), overall survival (OS) and safety (NCI CTCAE v 4.0).

Statistical methods: The PFS curve was estimated using the Kaplan-Meier method for the largest population to be analyzed. The confidence interval method was used as the criterion for the main analysis. OS was calculated in the same way as the secondary endpoint. Descriptive statistics will be used to analyze ORR, DCR, etc. It is expected that almonertinib plus anlotinib as first-line treatment will prolong median PFS and OS of advanced non-small cell lung cancer with EGFR sensitive mutation and TP53 mutation patients.

DETAILED DESCRIPTION:
Lung cancer is the most common solid tumor and the leading cause of cancer-related death in the world [1]. According to the Globocan analysis report of global cancer epidemic statistics in 2023, the number of new cases of lung cancer in the world reached 238,400, and the number of deaths reached 127,100, ranking first in all cancers [2]. There are about 815,000 new cases and 715,000 deaths in China every year, accounting for 23.8% of the total cancer deaths [1]. Non-small Cell Lung Cancer (NSCLC) is the most common pathological type of lung cancer, accounting for about 85% of all lung cancers [3]. About 70% of patients are locally advanced or advanced at the time of diagnosis, and only 25% of patients with NSCLC survive for more than 5 years after diagnosis. When patients receive traditional cytotoxic chemotherapy regimens, the 5-year relative survival rate of patients with advanced NSCLC is only 6%[4-6]. However, with the application of targeted therapy and immunotherapy in recent years, the 5-year survival rate of NSCLC patients receiving immunotherapy or targeted therapy can reach 15% to 50%[7-10].

EGFR mutation is one of the most common mutations in NSCLC, especially in lung adenocarcinoma.Since 2014, EGFR-TKI has become the standard first-line treatment for NSCLC patients with EGFR classical mutations.For advanced NSCLC patients with EGFR sensitive mutations and TP53 mutations, the benefit of single drug may be limited. Combination therapy may improve the survival and quality of life of advanced NSCLC patients with EGFR sensitive mutations and TP53 co-mutations, but there is still a lack of sufficient clinical trials to verify.

Almonertinib is a novel irreversible third-generation TKI. It is used for the treatment of adult patients with locally advanced or metastatic NSCLC with T790M mutation positive after prior EGFR-TKI treatment. The AENEAS study [25] is a multicenter, randomized, controlled, double-blind, phase III clinical trial comparing the efficacy and safety of almonertinib and gefitinib as first-line treatment for patients with locally advanced or metastatic NSCLC with EGFR19Del or L858R mutation. 429 untreated patients with locally advanced or metastatic disease harboring the EGFR19Del or L858R mutation were randomized to receive almonertinib at a dose of 110mg daily (n=214) or gefitinib at a dose of 250mg daily (n=215). The primary endpoint was investigator-assessed progression-free survival (PFS). Secondary endpoints included overall survival (OS), objective response rate (ORR), duration of response (DoR), and disease control rate (DCR). The results showed that the mPFS of almonertinib group and gefitinib group were 19.3 months and 9.9 months, ORR were 73.8% and 72.1%, DCR were 93.0% and 96.7%, DOR were 18.1 months and 8.3 months. Based on this study, on December 16, 2021, the NMPA officially approved almonertinib for the first-line treatment of adult patients with locally advanced or metastatic NSCLC with EGFR19Del or exon 21 L858R mutation.

Anlotinib is a novel multi-target oral tyrosine kinase inhibitor developed by China. It can effectively inhibit VEGFR, PDGFR, FGFR, PDGFRα and β and stem cell growth factor receptor (c-Kit) and other kinases, so it can play an effective role in anti-tumor angiogenesis and inhibition of tumor cell growth [29, 30]. A number of clinical trials have confirmed the significant efficacy of anlotinib in patients with advanced NSCLC. ALTER-0303 trial [31] was a randomized, double-blind, multicenter, controlled phase III clinical trial of anlotinib as a third-line or longer treatment for advanced NSCLC patients. A total of 437 subjects were enrolled in the study and randomly assigned to anlotinib group (n=294) and placebo group (n=143) at a ratio of 2:1. The primary endpoint was overall survival (OS). The secondary endpoints were PFS, ORR, DCR, Quality of Life (QoL), and safety. The results showed that anlotinib was superior to placebo in terms of OS and PFS. The median OS (mOS) and mPFS were 9.6 and 5.4 months, respectively, in the anlotinib group, and 6.3 and 1.4 months, respectively, in the placebo group. Meanwhile, the results of exploratory subgroup analysis showed that advanced NSCLC with EGFR mutation or EGFR wild type could benefit from clinical treatment in terms of OS and PFS. Based on this experimental result, on May 8, 2018, the China Food and Drug Administration (CFDA) officially approved single-agent anlotinib for the third-line and beyond treatment of advanced NSCLC patients.

To evaluate the efficacy and safety of almonertinib plus anlotinib as first-line treatment for advanced non-small cell lung cancer with EGFR sensitive mutation and TP53 mutation.

This study is an exploratory single-arm study. The specific treatment regimen is as follows: Non-squamous NSCLC: almonertinib (110 mg/d) plus anlotinib (12mg/d) is started on the first day of each treatment cycle and administered every three weeks until disease progression or intolerable toxicity. Anlotinib was given for two weeks, followed by one week off.

Patients are assessed for measurable disease at baseline, 6 weeks, 12 weeks after starting treatment, and every 9 weeks thereafter according to RECIST 1.1 criteria during the treatment period until disease progression or intolerable toxicity withdrawal. Following discontinuation of treatment, subjects are followed for survival status every 3 months until death. Subject safety was assessed during treatment according to NCI CTCAE Version 4.0 criteria. Subjects who experience an AE should be followed until the AE returns to baseline. The primary endpoints is Progression-free survival (PFS) . Secondary endpoints include objective response rate (ORR), overall survival (OS) and safety (NCI CTCAE v 4.0).

Statistical methods: The PFS curve was estimated using the Kaplan-Meier method for the largest population to be analyzed. The confidence interval method was used as the criterion for the main analysis. OS was calculated in the same way as the secondary endpoint. Descriptive statistics will be used to analyze ORR, DCR, etc. It is expected that almonertinib plus anlotinib as first-line treatment will prolong median PFS and OS of advanced non-small cell lung cancer with EGFR sensitive mutation and TP53 mutation patients.

ELIGIBILITY:
Inclusion Criteria:

Metastatic Non-squamous NSCLC is histologically or cytologically proven to be inoperable and cannot receive radical concurrent chemoradiotherapy. The conventional TNM stage was identified as stage IIIa-Ⅳb according to the International Association for the Study of Lung Cancer and the American Joint Committee on the Classification of Cancer 8th edition TNM Staging of Lung Cancer.

Patients with EGFR mutation and TP53 mutation advanced Non-squamous NSCLC. Patients who had not previously received systemic radiotherapy and chemotherapy or who had relapsed for more than 6 months of follow-up after onset of adjuvant chemotherapy.

At least one measurable lesion as determined by RECIST criteria. Male or female patients, age: 18-75 years of age. Performance score 0-1 based on Eastern Cooperative Oncology Group (ECOG) test. Expected survival period ≥12 weeks. Serum absolute number of neutrophils≥ 1.5 x 10^9/L, platelet ≥ 100 x10^9/L, and hemoglobin≥ 90g/L.

Serum bilirubin≤1.5 times ULNL, aspartate aminotransferase (AST) and adenosine triphosphate(ALT) ≤ 2.5 times ULN, alkaline phosphatase ≤ 5 times ULN.

Serum creatinine≤ the ULN or creatinine clearance ≥ 60 mL/min. Patients who had previously undergone surgery have recovered for more than 4 weeks from the beginning of the project.

Women with an intact uterus must have a negative pregnancy test within 28 days prior to enrolement in the study (unless it was 24 months after amenorrhea). If the pregnancy test is more than 7 days prior to initial dosing, a urine pregnancy test is required for verification (within 7 days prior to initial dosing).

If there is a risk of conception, all patients (whether male or female) are required to use contraceptive measures with an annual failure rate of less than 1% throughout the treatment period until 120 days after the last dose of the study drug.

Sign the inform consent form with good compliance.

Exclusion Criteria:

Those who are known to be allergic to the study drug almonertinib and anlotinib and its any components.

Intolerance to study drug treatment or allergy to the active ingredients or excipients of combined chemotherapy drugs.

Pregnancy or breastfeeding women or women who may be pregnant but are unwilling to take appropriate contraception.

Existing severe acute infections that are not under control; Or suppurative and chronic infections with delayed healing.

Pre-existing serious heart disease, including: congestive heart failure, uncontrolled high-risk arrhythmias, unstable angina pectoris, myocardial infarction, severe valvular heart disease, and refractory hypertension.

People suffering from uncontrollable neuropsychiatric diseases or mental disorders had poor compliance and were unable to cooperate and describe treatment responses; The conditions of patients with primary brain tumor or central nerve metastatic tumor were uncontrollable and the symptoms of cranial hypertension or neuropsychiatric were obvious.

Patients with hereditary bleeding tendency or coagulation dysfunction, or history of thrombosis or bleeding, and abnormal detection results of coagulation function related indicators.

Patients who are receiving thrombolytic or anticoagulant therapy due to high risk of thrombosis.

Patients with unhealed wounds, unhealed ulcers or unhealed fractures. Other conditions that the investigator considers to be inappropriate for the patient to participate in this trial.

Currently participating in interventional clinical research treatment, or have received other investigational drugs or used investigational device treatment within 4 weeks before the first dose.

Patients who have undergone major surgery within 4 weeks before the start of study treatment or are scheduled to undergo major surgery during the study period (except for surgery such as puncture or lymph node biopsy).

Pulmonary interstitial fibrosis with respiratory failure. Chronic obstructive pulmonary disease with respiratory failure. Active pulmonary tuberculosis; Active autoimmune disease requiring systemic therapy (such as the use of disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (such as thyroxine) is not considered systemic therapy; Those who are receiving systemic glucocorticoid therapy (excluding nasal spray, inhalation or other local glucocorticoids) or any other form of immunosuppressive therapy within 14 days before the first dose of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months]
  Progression-free survival

SECONDARY OUTCOMES:
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  overall survival
ORR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  objective response rate
DOR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Duration of Responst

CONTACTS AND LOCATIONS:
Overall Officials: Degan Lu, Principal Investigator — he First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital)
Locations (1):
- Degan Lu, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No